CLINICAL TRIAL: NCT02666963
Title: A Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of RTA 901 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 901-C-1503
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: RTA 901; RTA 901 capsules
MeSH Terms: interventions — ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RTA 901 10 mg or 40 mg or Placebo (Experimental): RTA 901 capsules (10 mg or 40 mg) or placebo taken orally in a single dose. Group 1: RTA 901 10 mg or matching placebo Group 2: RTA 901 20 mg or matching placebo Group 3: RTA 901 ≤ 40 mg or matching placebo Group 4: RTA 901 ≤ 80 mg or matching placebo Group 5: RTA 901 ≤ 160 mg or matching placebo Group 6: RTA 901 ≤ 320 mg or matching placebo Group 7: RTA 901 ≤ 640 mg or matching placebo Dose selection will be based on the safety, tolerability and available pharmacokinetics observed in prior study groups.
  Interventions: Drug: RTA 901 Capsules, 10 or 40 mg; Drug: Placebo
- RTA 901 Dose TBD or Placebo (Experimental): RTA 901 capsules, Dose TBD mg or placebo taken orally once daily for 14 days. Group 8: RTA 901 X mg or matching placebo Group 9: RTA 901 ≤Y mg or matching placebo Group 10: RTA 901 ≤Z mg or matching placebo The actual doses for Arm 2 will be selected based on the safety and available pharmacokinetic data obtained from Arm 1.
  Interventions: Drug: RTA 901 Capsules, 10 or 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: RTA 901 Capsules, 10 or 40 mg
Drug: Placebo

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetic profile of RTA 901 following escalating single and multiple oral doses of RTA 901 in healthy adult subjects.

This first-in-human, Phase 1, single-center study consists of single ascending doses (SAD) and multiple ascending doses (MAD) conducted in 2 parts. Part 1 (SAD) of this study will be conducted in approximately 56 healthy subjects in up to 7 groups. Each group will consist of up to 8 subjects who will be randomized in a 3:1 ratio to receive a single dose of RTA 901 or placebo, respectively. Safety, tolerability, and available pharmacokinetics through Day 4 will be assessed in each group prior to dose escalation.

Part 2 (MAD) of this study will be conducted in approximately 30 healthy subjects in up to 3 groups. Each group will consist of up to 10 subjects who will be randomized in a 4:1 ratio to receive 14 daily doses of RTA 901 or placebo, respectively. Safety, tolerability, and available pharmacokinetics through Day 17 will be assessed in each dosing group prior to dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age is between 18 and 55 years, inclusive.
* Women must be of non-childbearing potential and may not be pregnant, lactating, or breast-feeding. Non-childbearing potential is defined by at least one of the following criteria:

  1. At least 2 years spontaneous amenorrhea (not attributable to environmental or pathological causes, e.g., anorexia or excessive exercise) with follicle-stimulating hormone (FSH) in post-menopausal range at screening;
  2. At least 3 months post-surgical bilateral oophorectomy or tubal ligation; or
  3. Hysterectomy (must be greater than 5 years post-hysterectomy if due to cancer);
* Females must have negative results for pregnancy tests performed:

  1. At screening based on a urine specimen obtained within 28 days prior to initial study drug administration, and
  2. Prior to dosing based on a serum sample obtained on Day -1.
* If male, subject must be surgically sterile or practicing at least 1 of the following methods of contraception, from initial study drug administration through 90 days after administration of the last dose of study drug:

  1. Partner(s) using an IUD;
  2. Partner(s) using hormonal contraceptives (oral, vaginal, parenteral, or transdermal).
  3. Subject and/or partner(s) using double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jellies or creams);
  4. Total abstinence from sexual intercourse as the preferred life style of the subject; periodic abstinence is not acceptable.
* If male, subject agrees to abstain from sperm donation through 90 days after administration of the last dose of study drug.
* Body Mass Index (BMI) is ≥ 18 to < 32 kg/m2, inclusive.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the investigator.
* Must voluntarily sign and date each informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* History of clinically significant drug allergies, including allergies to any of the components of the investigational product and/or clinically significant food allergies as determined by the investigator; History of clinically significant drug allergies, including allergies to any of the components of the investigational product and/or clinically significant food allergies as determined by the investigator;
* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the investigator;
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* Requirement for any over-the-counter and/or prescription medication, vitamins, and/or herbal supplements on a regular basis.
* Use of any medications (over-the-counter and/or prescription medication), vitamins, and/or herbal supplements, within the 30-day period prior to study drug administration or within 5 half-lives (if known), whichever is longer.
* Recent (6-month) history of drug or alcohol abuse.
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab) at screening.
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days prior to study drug administration.
* Positive screen results for drugs of abuse, alcohol, or cotinine at screening or Day -1.
* Consumption of alcohol within 72 hours prior to study drug administration.
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, or Seville oranges within the 72-hour period prior to study drug administration.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
* Current enrollment in another clinical study.
* Previous enrollment in this study.
* Screening laboratory analyses that show any of the following abnormal laboratory results:

  1. Alanine transaminase (ALT) level above 1.2× the upper limit of normal (ULN).
  2. Aspartate transaminase (AST) level above 1.2× the ULN.
  3. Any other laboratory results that are outside of the laboratory normal reference range and considered clinically significant by the investigator.
* Clinically-significant abnormal ECG; ECG with QTc using Fridericia's correction formula (QTcF) > 450 msec is exclusionary.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive RTA 901.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by monitoring adverse events, physical examinations, clinical laboratory tests, 12-lead ECGs, and vital signs | 14 days
  Safety and tolerability will be assessed by monitoring adverse events, physical examinations, clinical laboratory tests, 12-lead ECGs, and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/